CLINICAL TRIAL: NCT04707326
Title: Defining the Potency of DTG/3TC for Suppressed HIV Patients in Real-life: the DUALING Study.
Acronym: DUALING
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other); Haaglanden Medical Centre (Other); Catharina Ziekenhuis Eindhoven (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Rijnstate Hospital (Other); Admiraal de Ruyter Hospital (Other); Spaarne Gasthuis (Other); Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, Casper Rokx, MD PhD, Erasmus Medical Center
Other Study IDs: DUALING
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- DTG based switchers to DTG/3TC: HIVRNA suppressed HIV patients who switched to DTG/3TC
- DTG based triple drug cART: Matched HIVRNA suppressed patients who remained on triple drug DTG based cART
- non-DTG based switchers to DTG/3TC
  Interventions: Drug: Dolutegravir / Lamivudine Pill
- non-DTG based triple drug cART: Matched HIVRNA suppressed patients who remained on triple drug non-DTG based cART

INTERVENTIONS:
Drug: Dolutegravir / Lamivudine Pill — HIVRNA suppressed patients without documented M184V mutation in HIV RT and who are hepatitis B immune or have no risk factors for acquiring hepatitis B
  Groups: non-DTG based switchers to DTG/3TC

SUMMARY:
This study aims to determine real-life clinical efficacy of virally suppressed patienst switching to DTG/3TC compared to DTG triple drug cART controls

DETAILED DESCRIPTION:
Dolutegravir (DTG) based dual antiretroviral therapy constitutes a paradigm shift from triple drug based therapy. Data outside clinical trials are scarce. This study evaluates the value of DTG/3TC in real life.

ELIGIBILITY:
Inclusion Criteria:

Plasma HIVRNA <50c/mL on triple drug cART regimen including 2NRTI In care in a HIV treatment center in the Netherlands Consented to ATHENA participation

Exclusion Criteria:

Documented mutations associated with 3TC or DTG resistance of at least low level Documented inadherence by the treating physician or HepB coinfection (cases only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible as case in the study, plasma HIVRNA must be <50c/mL on triple drug cART containing 2NRTI at switch to DTG/3TC and no key mutations associated with major 3TC (i.e. M184V/I only) or DTG resistance of at least low level according to the Stanford HIV drug resistance database should be present. Patients with no genotyping results available at baseline will be eligible for inclusion in this study. Cases should not have documented inadherence in the preceding 3 months or HepB coinfections. These data on adherence and HepB is routinely collected at switching to DTG/3TC. Controls are matched on predefined criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2040 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2026-11-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (9):
- Netherlands (9):
  - Rijnstate Hospital, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Spaarne Gasthuis, Haarlem
  - Erasmus MC, Rotterdam
  - MC Haaglanden, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Elisabeth Tweesteden Hospital, Tilburg

IPD SHARING:
Plan to Share IPD: Yes
Other research groups can contact the PI with a research question to obtain IPD.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Up to 15 years

REFERENCES:
- [Derived] Vasylyev M, Wit FWNM, Jordans CCE, Soetekouw R, van Lelyveld SFL, Kootstra GJ, Delsing CE, Ammerlaan HSM, van Kasteren MEE, Brouwer AE, Leyten EMS, Claassen MAA, Hassing RJ, den Hollander JG, van den Berge M, Roukens AHE, Bierman WFW, Groeneveld PHP, Lowe SH, van Welzen BJ, Richel O, Nellen JF, van den Berk GEL, van der Valk M, Rijnders BJA, Rokx C. Dolutegravir/Lamivudine Is Noninferior to Continuing Dolutegravir- and Non-Dolutegravir-Based Triple-Drug Antiretroviral Therapy in Virologically Suppressed People With Human Immunodeficiency Virus: DUALING Prospective Nationwide Matched Cohort Study. Open Forum Infect Dis. 2024 Mar 18;11(4):ofae160. doi: 10.1093/ofid/ofae160. eCollection 2024 Apr. PMID 38567196

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DTG Based Switchers to DTG/3TC | DTG Based Triple Drug cART | Non-DTG Based Switchers to DTG/3TC | Non-DTG Based Triple Drug cART
Started | 390 | 780 | 290 | 580
Completed | 390 | 780 | 290 | 580
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG Based Switchers to DTG/3TC | DTG Based Triple Drug cART | Non-DTG Based Switchers to DTG/3TC | Non-DTG Based Triple Drug cART | Total
Number analyzed (Participants) | 390 | 780 | 290 | 580 | 2040
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [37 to 57] | 48 [38 to 57] | 50 [39 to 59] | 50 [40 to 59] | 49 [38 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 92 | 61 | 122 | 321
  Male | 344 | 688 | 229 | 458 | 1719
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 100 | 35 | 79 | 248
  Not Hispanic or Latino | 356 | 680 | 255 | 501 | 1792
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
CD4 count nadir [Median (Inter-Quartile Range); unit: cells/mcL] | 330 [200 to 485] | 310 [190 to 471] | 290 [180 to 437] | 270 [170 to 380] | 300 [190 to 450]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy On Treatment (OT)
Description: Proportion of subjects with treatment failure in the DTG/3TC versus 3-drug DTG containing cART group up to 1 year of follow up in the on treatment population
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Based Switchers to DTG/3TC | DTG Based Triple Drug cART | Non-DTG Based Switchers to DTG/3TC | Non-DTG Based Triple Drug cART
Number analyzed (Participants) | 361 | 628 | 260 | 506
Participants | 5 | 5 | 2 | 4

2. Primary Outcome: Efficacy Intention to Treat (ITT)
Description: Proportion of subjects with treatment failure in the DTG/3TC versus 3-drug DTG containing cART group up to 1 year of follow up in the intention to treat population.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Based Switchers to DTG/3TC | DTG Based Triple Drug cART | Non-DTG Based Switchers to DTG/3TC | Non-DTG Based Triple Drug cART
Number analyzed (Participants) | 390 | 780 | 290 | 580
Participants | 34 | 89 | 32 | 73

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DTG Based Switchers to DTG/3TC | DTG Based Triple Drug cART | Non-DTG Based Switchers to DTG/3TC | Non-DTG Based Triple Drug cART
All-Cause Mortality (participants affected / at risk) | 0/390 | 0/780 | 0/290 | 0/580
Serious Adverse Events (participants affected / at risk) | 0/390 | 0/780 | 0/290 | 0/580
Other Adverse Events (participants affected / at risk) | 0/390 | 0/780 | 0/290 | 0/580

LIMITATIONS AND CAVEATS:
All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were collected during this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT04707326/Prot_SAP_000.pdf